CLINICAL TRIAL: NCT06657053
Title: Facteurs De Risques De Récidive D'épistaxis Chez L'adulte
Brief Title: Risk Factors of Epistaxis Recurrence in Adults
Acronym: FREA
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: EssaiClinique_FREA
Record Dates: First submitted 2024-10-22; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Epistaxis
Keywords: Risk Factors; Recurrent Epistaxis
MeSH Terms: conditions — Epistaxis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patient with nose bleeding: Evaluation of recurrence epistaxis during the year after a first episode

SUMMARY:
We study all patients admitted to the Emergency Department in the Institution between 01/2022 and 07/2023. The information about the recurrence of nose bleeding was searched on their medical file and by calling the patient to confirm ou get the information. Thus, several potentiel risk factors were studied.

The relation between recurrence and those factors were studied at first individually and then all the significant ones were analyzed with a multivarious statistical test.

DETAILED DESCRIPTION:
We study all patients admitted to the Emergency Department in the Institution between 01/2022 and 07/2023. The information about the recurrence of nose bleeding was searched on their medical file and by calling the patient to confirm ou get the information. Thus, several potentiel risk factors were studied : oral anticoagulants, sex, INR, anti-platelets drugs, diabetes, obesity, arterial hypertension, heart failure, hemoglobin at the admission, history of chronic rhinosinusitis, appointment with an ENT during the acute bleeding, sleep apnea, age, anatomic abnormality, recent surgery within 2 months, previous admission within 30 days in the emergency department, nasal trauma.

The relation between recurrence and those factors were studied at first individually and then all the significant ones were analyzed with a multivarious statistical test.

This study aim to provide a pronostic score of recurrence that can happen after the 3 fisrt weeks after the event. When a recurrence happens before 3 weeks, this was considered to be a non control of the bleeding episode.

This score will be then tested on our cohort to evaluate specificity and sensibility.

ELIGIBILITY:
Inclusion Criteria:

* Patient who is admitted at the emergency department between 01/2022 and 07/2023 for nose bleeding.
* Age over 18 yo

Exclusion Criteria:

* Opposition to be included
* Patient who has not his willness to provide opposition to participate.opposition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patientswho are admitted at the emergency department between 01/2022 and 07/2023
Sampling Method: Non-Probability Sample
Enrollment: 145 (Estimated)
Dates: Start 2024-11-02 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Survival without bleeding | 1 year
  Measuring the delay between the first epistaxis and a recurrence.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Grenoble Alpes, La Tronche, ISERE, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Addison A, Paul C, Kuo R, Lamyman A, Martinez-Devesa P, Hettige R. Recurrent epistaxis: predicting risk of 30-day readmission, derivation and validation of RHINO-ooze score. Rhinology. 2017 Jun 1;55(2):99-105. doi: 10.4193/Rhin16.259. PMID 28434017
- [Background] Abrich V, Brozek A, Boyle TR, Chyou PH, Yale SH. Risk factors for recurrent spontaneous epistaxis. Mayo Clin Proc. 2014 Dec;89(12):1636-43. doi: 10.1016/j.mayocp.2014.09.009. Epub 2014 Nov 6. PMID 25458126
- [Background] Chaaban MR, Zhang D, Resto V, Goodwin JS. Factors influencing recurrent emergency department visits for epistaxis in the elderly. Auris Nasus Larynx. 2018 Aug;45(4):760-764. doi: 10.1016/j.anl.2017.11.010. Epub 2017 Dec 6. PMID 29208334
- [Background] Melia L, McGarry GW. Epistaxis: update on management. Curr Opin Otolaryngol Head Neck Surg. 2011 Feb;19(1):30-5. doi: 10.1097/MOO.0b013e328341e1e9. PMID 21150620
- [Background] Pino Rivero V, Trinidad Ruiz G, Gonzalez Palomino A, Pardo Romero G, Pantoja Hernandez CG, Marcos Garcia M, Keituqwa Yanez T, Blasco Huelva A. [Considerations about ENT emergencies. Analysis of 30000 patients assisted in 10 years]. Acta Otorrinolaringol Esp. 2005 May;56(5):198-201. doi: 10.1016/s0001-6519(05)78600-3. Spanish. PMID 15960122
- [Background] Pallin DJ, Chng YM, McKay MP, Emond JA, Pelletier AJ, Camargo CA Jr. Epidemiology of epistaxis in US emergency departments, 1992 to 2001. Ann Emerg Med. 2005 Jul;46(1):77-81. doi: 10.1016/j.annemergmed.2004.12.014. PMID 15988431
- [Background] Tunkel DE, Anne S, Payne SC, Ishman SL, Rosenfeld RM, Abramson PJ, Alikhaani JD, Benoit MM, Bercovitz RS, Brown MD, Chernobilsky B, Feldstein DA, Hackell JM, Holbrook EH, Holdsworth SM, Lin KW, Lind MM, Poetker DM, Riley CA, Schneider JS, Seidman MD, Vadlamudi V, Valdez TA, Nnacheta LC, Monjur TM. Clinical Practice Guideline: Nosebleed (Epistaxis). Otolaryngol Head Neck Surg. 2020 Jan;162(1_suppl):S1-S38. doi: 10.1177/0194599819890327. PMID 31910111
- [Background] Cohen O, Shoffel-Havakuk H, Warman M, Tzelnick S, Haimovich Y, Kohlberg GD, Halperin D, Lahav Y. Early and Late Recurrent Epistaxis Admissions: Patterns of Incidence and Risk Factors. Otolaryngol Head Neck Surg. 2017 Sep;157(3):424-431. doi: 10.1177/0194599817705619. Epub 2017 May 2. PMID 28463569